CLINICAL TRIAL: NCT02406521
Title: Phase I Study of Radium-223 and Vascular Endothelial Growth Factor-Targeted Therapy in Patients With Metastatic Renal Cell Carcinoma and Bone Metastases
Brief Title: Exploratory Study of Radium-223 and VEGF-Targeted Therapy in Patients With Metastatic Renal Cell Carcinoma and Bone Mets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Mark Pomerantz, MD, Assistant Professor of Medicine, Harvard Medical School, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-523
Record Dates: First submitted 2015-03-16; First posted 2015-04-02 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: Metastatic renal cell carcinoma; mRCC
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — pazopanib; Sorafenib; Radium-223; radium Ra 223 dichloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: Pazopanib with Radium-223 (Experimental): No prior targeted therapy
  * Pazopanib oral, daily and at predetermined dosage per cycle
  * Radium-223 predetermined dosage via IV, per cycle
  Interventions: Drug: Pazopanib; Drug: Radium-223
- Arm B: Sorafenib with Radium-223 (Experimental): At least one line of prior targeted therapy:
  * Sorafenib at predetermined dosage, mouth twice daily
  * Radium-223 predetermined dosage via IV, per cycle
  Interventions: Drug: Sorafenib; Drug: Radium-223

INTERVENTIONS:
Drug: Pazopanib
  Other Names: Votrient
  Arms: Arm A: Pazopanib with Radium-223
Drug: Sorafenib
  Other Names: Nexavar®
  Arms: Arm B: Sorafenib with Radium-223
Drug: Radium-223
  Other Names: Radium 223 Dichloride; Xofigo®

SUMMARY:
This research study is comparing different drug combinations as a possible treatment for metastatic renal cell carcinoma (mRCC) and bone metastases.

The names of the study interventions involved in this study are:

* Combination of Radium-223 and Sorafenib
* Combination of Radium-223 and Pazopanib

DETAILED DESCRIPTION:
The FDA (the U.S. Food and Drug Administration) has not approved the combination of sorafenib and radium-223 or the combination of pazopanib and radium-223 as a treatment for any disease. Sorafenib and pazopanib are both approved as single agents for the treatment of metastatic renal cell carcinoma. Additionally, radium-223 is FDA approved for the treatment of advanced prostate cancer and has shown to have effects on prostate cancer.

Currently, there are limited options for patients with metastatic renal cell cancer who also have bone metastases. Bone metastases are related to a higher incidence of skeletal complications, including skeletal pain, fractures, spinal cord compression, and an increase in the amount of calcium in blood. Such skeletal complications could result in radiation or surgery to the bone. Since radium-223 is shown to be effective for patients with metastatic prostate cancer who also have bone metastases, researchers want to explore radium-223 with VEGF-targeting therapies to understand how the drug combinations affect safety, quality of life, incidence of skeletal complications, and the progression of cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Documented pathologic diagnosis of RCC. All subtypes eligible including but not limited to clear cell, papillary, chromophobe, collecting duct carcinoma, medullary carcinoma, and unclassified categories. Sarcomatoid and rhabdoid differentiation are allowed.
* Presence of at least one metastatic bone lesion(s). Patients with non-measurable bone-only disease are allowed.
* ECOG performance status of 0-2 (Appendix A).
* Must have adequate organ and bone marrow function.

  * Absolute neutrophil count (ANC) ≥ 1500/mm3 (without use of G-CSF 4 weeks prior to enrollment).
  * Platelet count ≥100,000/mm3.
  * Hemoglobin ≥ 9 g/dL (transfusions allowed).
  * ALT and AST ≤ 3.0 x the upper limit of normal (ULN).
  * Total bilirubin ≤ 1.5 x ULN. For participants with Gilbert's disease ≤ 3.0 mg/dL.
  * Calculated creatinine clearance ≥ 30 mL/min using the Cockroft-gault equation.
  * Urine protein-to-creatinine (UPC) ratio ≤ 2 mg/mg creatinine or 24-hour urine protein < 2 g.
* Recovery to baseline or ≤ grade 1 CTCAE version 4.0 from toxicities related to any prior treatment, unless adverse events are clinically non-significant and/or stable on supportive therapy.
* Capable of understanding and complying with the protocol requirements and has signed the informed consent document.
* Sexually active participants and their partners must agree to use medically accepted methods of contraception.
* Female participants of childbearing potential must not be pregnant at screening.
* Sexually active participants (men and women) must agree to use highly effective contraceptive methods during the course of the study and for 6 months after completing treatment with radium-223.

Exclusion Criteria:

* For patients in the sorafenib cohort, no prior therapy with sorafenib is allowed and at least 1 line of prior therapy is required including prior: VEGF-targeting therapy (such as sunitinib, axitinib, tivozanib, bevacizumab), mTOR-targeting therapy (such as everolimus, temsirolimus), immunotherapy (such as anti-PD-1 or anti-PD-L1), cytokine therapy (such as interleukin-2, IFN-a) or cytotoxic systemic chemotherapy allowed.
* For patients in the pazopanib cohort, no prior systemic therapy for mRCC is allowed, with the exception of prior cytokine therapy (such as interleukin-2, IFN-a), immunotherapy (such as anti-PD-1 or anti-PD-L1), or supportive therapies (such as zoledronic acid, denosumab).
* Receipt of any type of small molecular kinase inhibitor (including investigational kinase inhibitors) within 2 weeks of enrollment or receipt of any anti-cancer therapy (including investigational therapy, monoclonal antibodies, cytokine therapy) within 3 weeks of enrollment.
* Radiation therapy for bone metastases within 2 weeks, other external radiation therapy within 4 weeks of enrollment.
* Received prior hemibody external radiotherapy.
* Prior therapy with radium-223 or systemic radiotherapy (such as samarium, strontium).
* Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy, radiosurgery, or surgery and stable for at least 4 weeks of enrollment as documented by MRI or CT imaging. Treated brain metastases are defined as having no ongoing requirement for steroids (must be off steroids for at least 4 weeks) and no evidence of progression or hemorrhage after treatment for at least 4 weeks of enrollment as documented by MRI or CT imaging.
* Imminent or established spinal cord compression based on clinical and/or imaging. In patients with untreated imminent or established spinal cord compression, treatment with standard of care as clinically indicated should be completed at least 4 weeks before enrollment.
* The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:

  * Cardiovascular disorders:

    * Symptomatic congestive heart failure, unstable angina pectoris, serious cardiac arrhythmias.
    * uncontrolled hypertension defined as sustained BP > 150 mm Hg systolic or > 100 mm Hg diastolic despite optimal antihypertensive treatment.
    * Stroke (including transient ischemic attack), myocardial infarction, or other ischemic event within 12 weeks of enrollment.
    * Thromboembolic event (such as deep venous thrombosis, pulmonary embolism) within 4 weeks of enrollment.
  * GI disorders including those associated with a high risk of perforation or fistula formation:

    * Tumors invading the GI-tract, active peptic ulcer disease, inflammatory bowel disease, diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis or acute obstruction of the pancreatic or biliary duct, or gastric outlet obstruction.
    * Abdominal fistula, gastrointestinal perforation, bowel obstruction, or intraabdominal abscess within 12 weeks before enrollment. Note: Complete healing of an intra-abdominal abscess must be confirmed before enrollment.
  * Clinically significant hematuria, hematemesis, or hemoptysis of > 0.5 teaspoon (2.5 ml) of red blood, or other history of significant bleeding (such as pulmonary hemorrhage) within 4 weeks of enrollment.
  * Other clinically significant disorders such as:

    * Active infection requiring systemic treatment, infection with human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness, or chronic hepatitis B or C infection.
    * Serious non-healing wound or ulcer.
    * Malabsorption syndrome.
    * Symptomatic hypothyroidism.
    * Moderate to severe hepatic impairment (Child-Pugh B or C).
    * Requirement for hemodialysis or peritoneal dialysis.
    * History of solid organ transplantation.
  * Major surgery (such as GI surgery) within 6 weeks of enrollment. However, subjects who have had a nephrectomy may be enrolled 4 weeks after surgery, providing there are no wound-healing complications. Subjects with clinically relevant ongoing complications from prior surgery are not eligible. The following are not considered to be major procedures: Thoracentesis, paracentesis, port placement, laparoscopy, thoracoscopy, bronchoscopy, endoscopic ultrasonographic procedures, mediastinoscopy, skin biopsies, incisional biopsies, imaging-guided biopsy for diagnostic purposes, and routine dental procedures.
  * QTcF > 470 msec within 4 weeks of enrollment. If the initial QTcF is found to be > 470 ms, two additional EKGs separated by at least 3 minutes should be performed. If the average of these three consecutive results for QTcF is ≤ 470 ms, the subject meets eligibility in this regard.
  * Pregnant or lactating females.
  * Inability to swallow tablets or capsules.
  * Previously identified allergy or hypersensitivity to components of the study treatment formulations.
  * Diagnosis of another malignancy within 2 years of enrollment, except for superficial skin cancers, or localized, low grade tumors deemed cured and not treated with systemic therapy by the principal investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-04; Primary Completion 2017-12 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Biomarkers of osteoblast and osteoclast activity | Baseline, 2 Years

SECONDARY OUTCOMES:
Symptomatic skeletal events (SSEs) | Baseline, 2 Years
Time to SSE | Baseline, 2 Years
Quality of life using the FKSI-19 | Baseline, 2 Years
Pain using the Brief Pain Inventory (Short Form) | Baseline, 2 Years
Analgesic use | Baseline, 2 Years
Overall response rate by RECIST version 1.1 | 2 Years
Duration of response by RECIST version 1.1 | 2 Years
Overall survival | 2 Years
Progression-free survival | 2 Years
Response as determined by PERCIST Criteria | 2 Years
Response as determined by MDA Bone Response Criteria | 2 Years
Response within bone biomarker subgroups | 2 Years
Time to first SSE within bone biomarker subgroups | 2 Years
PFS within bone biomarker subgroups | 2 Years
OS within bone biomarker subgroups | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Mark Pomerantz, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No